## STATISTICAL ANALYSIS PLAN: INDV-6000-405 Addendum

**Protocol Title:** A Single-Dose Study to Evaluate the Relative Bioavailability, Safety, and Tolerability of SUBLOCADE at Alternative Injection Locations in Adults

Final Version: 19 Mar 2024

**NCT:** NCT05704543

## Statistical Analysis Plan Addendum

Protocol ID: INDV-6000-405

Date: 19MAR2024

## **Description:**

After database lock, it was noted that the appendix of the SAP the following definition was used to derive medications prior to SUBLOCADE injection.

| | Start Date of Non-Study Medication | | |
|---|---|---|---|
| End Date of Non-<br>Study Medication | Missing | < Start date of SUBOXONE | ≥ Start date of SUBOXONE<br>and ≤ end date of<br>SUBOXONE |
| Missing (includes flagged as "Ongoing") | Prior<br>Concomitant<br>(Run-In) | Prior<br>Concomitant (Run-<br>In) | Concomitant (Run-In) |
| < Start date of SUBOXONE | Prior | Prior | Data Error |
| ≥ Start date of<br>SUBOXONE and ≤<br>end date of<br>SUBOXONE | Prior<br>Concomitant<br>(Run-In) | Prior<br>Concomitant (Run-<br>In) | Concomitant (Run-In) |

However, in the last row of this table, it implies that prior medications and Run-In concomitant medications do not include a medication started before injection and ended after last dose of SUBOXONE. The first column last row should not include the clause "and ≤ end date of SUBOXONE".

In addition, medications should be considered run-in concomitant as long as its start date is between start of SUBOXONE and SUBLOCADE injection date (if injection took place). Therefore, the last column should be split into two situations, with and without injection.

After modification, the definition should read the following:

| | Start Date of Non-Study Medication | | | |
|---|---|---|---|---|
| End Date of<br>Non-Study<br>Medication | Missing | < Start date of SUBOXONE | ≥ Start date of<br>SUBOXONE if no<br>injection | ≥ Start date of<br>SUBOXONE and ≤<br>SUBLOCADE<br>injection date if there<br>is SUBLOCADE<br>injection |
| Missing<br>(includes<br>flagged as<br>"Ongoing") | Prior<br>Concomitant<br>(Run-In) | Prior<br>Concomitant<br>(Run-In) | Concomitant (Run-In) | Concomitant (Run-In) |
| < Start date of SUBOXONE | Prior | Prior | Data Error | Data Error |

| ≥ Start date of<br>SUBOXONE | Prior<br>Concomitant<br>(Run-In) | Prior<br>Concomitant<br>(Run-In) | Concomitant (Run-In) | Concomitant (Run-In) |
|---|---|---|---|---|
|---|---|---|---|---|

## Implications:

Run-In concomitant medications flag and consequently, Table 14.1.5.2 will be updated.